CLINICAL TRIAL: NCT06308744
Title: Self-administered Mindfulness Interventions Reduce Stress in a Large, Randomized Controlled Multi-site Study
Brief Title: A Large Multi-site Study on Self-administered Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: University Grenoble Alps (Other); University of Utah (Other); Seeburg University (Unknown); Ludwig-Maximilians - University of Munich (Other); University of Houston (Other); Loyola Marymount University (Other); Ashland University (Unknown); The College at Brockport (Other); Medical University of South Carolina (Other); Australian National University (Other); The University of Queensland (Other); University of North Florida (Other); University of Wuerzburg (Other); Iowa State University (Other); Goldsmiths, University of London (Other); Pennsylvania Western University (Unknown); University of Konstanz (Other); Springfield College (Other); Glendale Community College (Unknown); St. Olaf College (Unknown); University of Limerick (Other); Northumbria University (Other); Wittenberg University Ohio (Unknown); University of Edinburgh (Other); University of California, Merced (Other); University of Southern Indiana (Unknown); Pace University (Other); Toronto Metropolitan University (Other); Wayne State University (Other); Memorial University of Newfoundland (Other); University College, London (Other); DigiPen Institute of Technology Redmond (Unknown); University of Canberra (Other); University of Northern Iowa (Other); Idaho State University (Other); Behavioural Science Institute (Other); Radboud University Medical Center (Other); Eastern Oregon University (Unknown); Charles University, Czech Republic (Other); University of Milano Bicocca (Other); Spiessens Coaching Solutions Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-5212-4387
Record Dates: First submitted 2024-02-27; First posted 2024-03-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Body Scan Meditation; Loving-Kindness Meditation; Mindful Breathing Meditation; Mindful Walking Meditation; Control Condition
Keywords: Mindfulness; self-administered mindfulness; self-help mindfulness; multi-site study; stress reduction

STUDY DESIGN:
Intervention Model Description: The current multi-site project followed the route of a parallel randomized controlled trial. Each participant was randomly allocated to either an experimental condition corresponding to a 15-minute audio listening of one of four different mindfulness exercises (i.e., mindful walking, mindful breathing, body scan and loving kindness meditation) or to a control condition (i.e., listening to a 15-minute audio story excerpt). Participants who were assigned to the control group randomly listened to an excerpt of one of the three stories that the investigators selected for the present study.
Who Masked: Participant
Masking Description: Participants were not aware of the experimental condition in which they were randomly allocated. Data collection was performed blind to the experimental conditions, but data analysis was not performed blind. However, given that all analyses were pre-registered, it is unlikely that the lack of blinding in data analysis introduced bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness conditions (Experimental): Participants will engage in a 15-minute mindfulness meditation session. Within this framework, four distinct experimental conditions will be introduced, each showcasing a unique mindfulness exercise: Body Scan, Mindful Breathing, Mindful Walking, and Loving-Kindness Meditation. The audio tracks of the mindfulness experimental conditions is embedded in the Qualtrics survey.
  Interventions: Behavioral: Body-scan meditation; Behavioral: Mindful Breathing meditation; Behavioral: Loving Kindness meditation; Behavioral: Mindful Walking
- Listening of a story (Active Comparator): Participants in the active control condition listened to a 15-minute story. The audio track of the control condition is embedded in the Qualtrics survey.
  Interventions: Behavioral: Listening of a story

INTERVENTIONS:
Behavioral: Body-scan meditation — Participants listen to a 15-minute Body-Scan mindfulness meditation recorded by a certified instructor. The audio track is embedded in the Qualtrics survey.
  Arms: Mindfulness conditions
Behavioral: Mindful Breathing meditation — Participants listen to a 15-minute Mindful Breathing mindfulness meditation recorded by a certified instructor. The audio track is embedded in the Qualtrics survey.
  Arms: Mindfulness conditions
Behavioral: Loving Kindness meditation — Participants listen to a 15-minute Loving Kindness mindfulness meditation recorded by a certified instructor. The audio track is embedded in the Qualtrics survey.
  Arms: Mindfulness conditions
Behavioral: Mindful Walking — Participants listen to a 15-minute Mindful Walking mindfulness meditation recorded by a certified instructor. The audio track is embedded in the Qualtrics survey.
  Arms: Mindfulness conditions
Behavioral: Listening of a story — Participants listen to a 15-minute story. The audio track is embedded in the Qualtrics survey.
  Arms: Listening of a story

SUMMARY:
The use of self-administered mindfulness interventions has increased in recent years. The effectiveness of these interventions on regulating stress/emotions, however, is debated. In the present multi-site study (Nsites = x, Nparticipants = x), the investigators aimed to investigate the effectiveness of four single, brief stand-alone mindfulness exercises in a population unfamiliar with mindfulness meditation. The investigators tested these four interventions in comparison to non-mindful active control conditions using an adaptive Bayesian design. The investigators found [evidence for the efficacy of x exercises/no evidence for the efficacy of x exercises] with an estimated mean effect size of [xx/xx]. This means that… or The investigators recommend that… [recommendation will be provided].

DETAILED DESCRIPTION:
Author's note:

The current project was pre-registered on the Open Science Framework (OSF) on March 22nd 2022, which was prior to the start of data collection (https://doi.org/10.17605/OSF.IO/UF4JZ). Data collection started on March 23th 2022 and ended on June 30th 2022. The investigators are retroactively registering the current study upon request of the editor who reviewed their manuscript (to comply with the editorial policies and formatting requirements of the target journal). The following protocol is an abbreviated version of the one the investigators uploaded on the OSF (https://osf.io/us5ae).

The upcoming multi-site project 'Self-administered mindfulness interventions reduce stress in a large, randomized controlled multi-site study' will aim to deliver in-depth insights into how self-administered mindfulness exercises impact stress reduction. It will focus on evaluating the effectiveness of self-administered mindfulness exercises in reducing stress among a large and diverse group of participants. Participants will be randomized to one of the audio-mindfulness exercises or to an active control condition. All exercises and the active control condition instructions will be designed to last 15 minutes. The active control condition will consist of a matched non-mindful listening condition in which mindfulness will not be mentioned. After the end of this intervention, a questionnaire will assess the self-reported stress of individuals with a short-term efficacy span. The study will also investigate the potential role of neuroticism as a moderator, as previous research has negatively associated neuroticism with mindfulness traits (i.e., the ability to be grounded in the present moment; Walsh et al., 2009). Bayesian sequential analysis tools (Schönbrodt et al., 2017) will be used to monitor the progress and to test the efficacy of each self-administered mindfulness exercise (i.e., upon reaching a predefined Bayes Factors). The results of this multi-site project will provide an answer to whether brief, stand-alone mindfulness exercises can demonstrate efficacy in decreasing levels of stress in individuals.

ELIGIBILITY:
* Inclusion Criteria:
* Adult participants aged 18 years or older at the time of the study.
* Participants who are English native speakers or who self-assessed their English language proficiency at the C1/C2 levels from the Common European Framework of Reference for Languages.
* Exclusion Criteria:
* Participants with a current or past history of mental illnesses (assessed via a pre-screening question).
* Participants who have engaged in meditation within six months prior to data collection.
* Participants who do not meet the English language proficiency requirements specified in the 'Inclusion Criteria' section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2239 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Stress | Day 1 - After the listening of the audio track, approximately 25 minutes after the beginning of the survey
  Participants answer the 20-item State-Trait Anxiety Inventory, Form Y-1 (STAI19). Participants indicate how they felt in that exact moment on 20 items (e.g., "I am tense"; "I feel frightened"; ωu = 0.92) on a 4-point scale (1 = Not at all, 2 = Somewhat, 3 = Moderately so, 4 = Very much so). By using the STAI Form Y-1 scale, the investigators aimed to measure the short-term effects of stress on individuals. This scale, after all, has been shown to correlate with biomarkers of stress in previous research (salivary α-amylase).

SECONDARY OUTCOMES:
Emotion dimensions | Day 1 - After the listening of the audio track, approximately 25 minutes after the beginning of the survey
  Participants filled in the Self-Assessment Manikin scale, a 3-item non-verbal pictorial assessment technique that measures emotions on three different dimensions, namely pleasure, arousal, and dominance. The Self-Assessment Manikin scale is the picture-oriented version of the widely used Semantic Differential Scale. This instrument measures the three-dimensional structure of stimuli, objects, and situations with 18 bipolar adjective pairs that can be rated along a 9-point scale. This measure was not the primary dependent variable of the study, but the investigators added it in the study for the exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sparacio, Ph.D., Principal Investigator — Swansea University & Universite Grenoble Alpes, A*STAR
Locations (1):
- Swansea University, Swansea, Wales, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan for IPD for the current study.

REFERENCES:
- [Derived] Sparacio A, IJzerman H, Ropovik I, Giorgini F, Spiessens C, Uchino BN, Landvatter J, Tacana T, Diller SJ, Derrick JL, Segundo J, Pierce JD, Ross RM, Francis Z, LaBoucane A, Ma-Kellams C, Ford MB, Schmidt K, Wong CC, Higgins WC, Stone BM, Stanley SK, Ribeiro G, Fuglestad PT, Jaklin V, Kubler A, Ziebell P, Jewell CL, Kovas Y, Allahghadri M, Fransham C, Baranski MF, Burgess H, Benz ABE, DeSousa M, Nylin CE, Brooks JC, Goldsmith CM, Benson JM, Griffin SM, Dunne S, Davis WE, Watermeyer TJ, Meese WB, Howell JL, Standiford Reyes L, Strickland MG, Dickerson SS, Pescatore S, Skakoon-Sparling S, Wunder ZI, Day MV, Brenton S, Linden AH, Hawk CE, O'Brien LV, Urgyen T, McDonald JS, van der Schans KL, Blocker H, Ng Tseung-Wong C, Jiga-Boy GM. Self-administered mindfulness interventions reduce stress in a large, randomized controlled multi-site study. Nat Hum Behav. 2024 Sep;8(9):1716-1725. doi: 10.1038/s41562-024-01907-7. Epub 2024 Jun 11. PMID 38862815

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT06308744/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT06308744/ICF_001.pdf